CLINICAL TRIAL: NCT01436721
Title: The Randomized Clinical Trial of Surgicel® Absorbable Haemostat Covering the Raw Cut Surface During the Hepatectomy
Brief Title: Use of an Oxidized Regenerated Cellulose After Hepatic Surgery
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jia Fan, Vice President of zhongshan hospital, Fudan University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCI-125-001
Record Dates: First submitted 2011-09-13; First posted 2011-09-20 (Estimated); Last update posted 2011-09-20 (Estimated); Status verified 2011-09

CONDITIONS: Liver Neoplasms
Keywords: Effectiveness; Device success; Hepatectomy
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Surgicel® absorbable Haemostat (No Intervention)
  Interventions: Device: Surgicel® absorbable Haemostat

INTERVENTIONS:
Device: Surgicel® absorbable Haemostat — The raw cut surface was covered with Surgicel® absorbable Haemostat or none but was dried by using fine sutures and an argon beam to achieve complete haemostasis.

SUMMARY:
Hepatectomy is one of the best treatments for malignant or benign lesions of the liver. The mortality and morbidity rates after hepatectomy have declined in recent years because of the precise measurement of liver functional reserve, a better understanding of liver anatomy, meticulous haemostasis during operation and improved postoperative management. Although surgical techniques have improved, life-threatening complications, such as intra-abdominal bleeding, bile leakage and subphrenic infection, now cannot be completed avoided. The local complications were most associated with the liver section treatment during the operation. Hence, the need for safer and more effective hemostatic treatment than the conventional approaches, such as intraoperative pressure by surgical gauze, ligatures, and electrocoagulation by mono- or bipolar instruments.

Surgicel® absorbable Haemostat is a sterile absorbable knitted fabric prepared by the controlled oxidation of regenerated cellulose. After Surgicel® has been saturated with blood, it swells into a brownish or black gelatinous mass which aids in the formation of a clot, thereby serving as a haemostatic adjunct in the control of local haemorrhage barriers on section.

The present randomized clinical trial was designed to evaluate the efficacy and safety of Surgicel® absorbable Haemostat covering the raw cut surface during the hepatectomy.

DETAILED DESCRIPTION:
This is a prospective, randomized, single-center investigation with a minimum of forty (40) controlled study subjects designed to evaluate the safety and effectiveness of the Surgicel® absorbable Haemostat as an absorbable hemostat in the hepatic surgical patient population.

Subjects who are undergoing hepatic surgical procedures should be considered for this investigation. The raw cut surface was covered with Surgicel® absorbable Haemostat or none but was dried by using fine sutures and an argon beam to achieve complete haemostasis. Subjects can be pre-screened utilizing standard of care data for the specified inclusion/exclusion criteria to ensure that they are eligible for treatment in the investigation. If the subject appears to qualify for the investigation, the subject will then be asked to give his/her written informed consent. All subjects will be followed through their hospitalization. Follow-up evaluations will include time to removal of wound drain, the amount of effusion, length of postoperative hospital stay, and incidence of postoperative morbidity.

From baseline to the final study exam, data pertaining to the investigational objectives will be recorded on the appropriate case report forms at the predetermined study intervals.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is 18 years to 70 Years
2. The subject is undergoing major hepatectomy (right hemihepatectomy, right posterior sectionectomy, and right anterior sectionectomy) without concomitant operation on another organ or anastomosis between bile ducts, or bile ducts and the digestive tract, and no abdominal infection
3. The subject is willing and able to provide appropriate informed consent
4. The subject is willing and able to comply with the requirements of the study protocol, including the predefined follow-up evaluations

Exclusion Criteria:

1. The subject is known or suspected to be pregnant (verified in a manner consistent with institution's standard of care), or is lactating
2. The subject has an active infection at the surgical site
3. The use of hemostatic agents are contraindicated for the subject
4. The subject has a known bleeding disorder (including thrombocytopenia [< 100,000 platelet count], thromboasthenia, hemophilia, or von Willebrand disease)
5. The subject has had surgery at the intended application site ≤ 6 months before the current surgical procedure
6. The subject is unavailable for follow-up
7. The subject is currently participating in another investigational device or drug trial
8. Administration of non-steroidal anti-inflammatory drugs (NSAIDs) or anti-platelet agents within 1 week before surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-08; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
the size of any subphrenic collection or pleural effusion | up time to the drainage tube removed, an expected average of 1 week
  If large amounts of ascites developed, diuretics were given and the volume of infusion was limited. Before removed grainage tube, all patients were examined by ultrasonography performed by a doctor without knowledge of the study. The size of any subphrenic collection or pleural effusion was recorded. The drainage tube was removed when the leakage per 24 h was less than 50 cm3, the appearance of the secretion had changed from hematic to serous, and no bilious or infectious discharge was present, as determined by observation.

SECONDARY OUTCOMES:
time to removal of wound drain | up time to removal of wound drain, an expected average of 1 week
length of postoperative hospital stay | up time to discharge from hospital,an expected average of 2 weeks
incidence of postoperative morbidity | up time to discharge from hospital,an expected average of 2 weeks
  After surgery, albumin, prophylactic broad-spectrum antibiotics, and enriched branched amino acid and fat emulsion (medium- and long-chain triglycerides), were given for 5-7 days until oral intake was possible.Ultrasonography-guided paracentesis or insertion of a second drainage tube was performed in patients with a subphrenic collection accompanied by fever (38.5◦C or higher) or a raised white blood cell count.

CONTACTS AND LOCATIONS:
Overall Officials: Jia Fan, MD, Principal Investigator — Liver cancer institute, fudan university
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China